CLINICAL TRIAL: NCT04913038
Title: Assessment of the Validity of the ANI in Children Over 2 Years of Age and Prepubescent Ventilated and Sedated in Pediatric Intensive Care.
Brief Title: Validation of the ANI in Perpubescent Patients in Pediatric Intensive Care Unit.
Acronym: ANI-EP
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_92; 2021-A00487-34 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-05-17; First posted 2021-06-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2023-11

CONDITIONS: Pain; Pediatric ALL
Keywords: Intensive Care Units,; Pain Measurement; ANI, Analgesia Nociception Index; Pediatric,
MeSH Terms: conditions — Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- case group: children over 2 years of age and prepubescent ventilated and sedated in pediatric intensive care.

SUMMARY:
The ANI monitor is a medical device allowing to measure the response of the autonomic nervous system to a painful stimulus.

In the pediatric population under general anesthesia, the ANI score can detect failure of locoregional anesthesia; ANI decreases after painful stimulation during surgery, more markedly with smaller doses of Remifentanil.

To date, measurement of ANI in sedated children in pediatric intensive care has not been performed or validated as a method of assessing pain and discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Prebubescent chilren (up to 2 years old) Admited in PICU Sedated, ventilated

Exclusion Criteria:

* Non sinusal rythm
* Atropine
* Pace-macker

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children over 2 years of age and prepubescent ventilated and sedated in pediatric intensive care
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Analgesia Nociception Index (ANI) minimum | at 10 minutes before the painful care
ANI minimum | at 30 minutes (average lenght of painful care)
ANI minimum | at 10 minutes after the painful care

SECONDARY OUTCOMES:
Variation of ANI minimum between before and after a painful care | From 10 minutes before the care to 10 minutes after the care
the correlation between ANI minimum and the COMFORT B behavioral scale. | From 10 minutes before the care to 10 minutes after the care
  The COMFORT BEHAVIOURAL (COMFORT-B) SCALE consists of six items: alertness, calmness, respiratory response, body movements, facial tension and muscle tone. Each item goes from 1 to 5, assessing the different intensities. The sum of the six ratings leads to a final score ranging from a minimum of 6 to a maximum of 30. A patient is considered to be under-sedated in case of COMFORT-B scores of 23 or higher, over-sedated in case of COMFORT-B scores of 10 or lower.
the ability of ANI minimum to distingush painful from non painful patient | From 10 minutes before the care to 10 minutes after the care
Area under the ROC curve of ANI min calculated over all measurements | From 10 minutes before the care to 10 minutes after the care

CONTACTS AND LOCATIONS:
Overall Officials: Morgan RECHER, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France

REFERENCES:
- [Derived] Barat A, Wojtanowski A, Behal H, Flocteil M, Leteurtre S, De Jonckheere J, Recher M. Evaluation of the Analgesia Nociception Index (ANI) as an indicator of discomfort in deeply sedated, prepubescent patients. J Clin Monit Comput. 2025 Sep 9. doi: 10.1007/s10877-025-01355-2. Online ahead of print. PMID 40924276